CLINICAL TRIAL: NCT00900458
Title: Adjustment of the Venous Reserve Capacity by Aerobic Exercise in Women at Increased Risk of Hypertensive Pregnancy Complications
Brief Title: Exercise Induced Improvement of the Venous Reserve Capacity in Formerly Pre-eclamptic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Ralph Scholten, Drs, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: exercise and pre-eclampsia
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Preeclampsia
Keywords: preeclampsia; low vs high plasma volume
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): formerly preeclamptic women with low plasma volume
  Interventions: Behavioral: Aerobic Exercise training
- 2 (Active Comparator): formerly preeclamptic women with normal plasma volume
  Interventions: Behavioral: Aerobic Exercise training
- 3 (Other): Healthy controls
  Interventions: Behavioral: Aerobic Exercise training

INTERVENTIONS:
Behavioral: Aerobic Exercise training — aerobic exercise training (cycling)

SUMMARY:
Primary objective:

* To investigate whether physical exercise prior to pregnancy in formerly preeclamptic women results in a comparable improvement of vascular and endothelial functioning as in women who had an uneventful pregnancy.

Secondary objectives:

* Which cardiovascular and endothelial parameters are involved in the vascular adaptation to training in women with a history of preeclampsia.
* To study the vascular adaptation in the (next) pregnancy in women with a history of preeclampsia compared with women with a history of an uncomplicated pregnancy, after improvement of their physical condition by exercise training.

This study is important in order to get a better understanding of the vascular and endothelial factors involved in preeclampsia and the effects of training on this profile. Results of this study can contribute to the improvement of preventing hypertensive complications in pregnancy and reduction of life time risk of cardiovascular disease in formerly preeclamptic women.

DETAILED DESCRIPTION:
In the Netherlands almost 15.000 women each year develop hypertensive complications like preeclampsia during their first pregnancy. In the western world these complications account for the most substantial attribution to neonatal and maternal morbidity and mortality. The exact etiology of this disease cascade is still unknown. There is accumulating evidence that subclinical abnormalities and preexistent haemodynamic, haemostatic and endothelial factors are involved, and thought to have negative impact on placental and endothelial functioning. The same factors are found to be risk factors for cardiovascular incidents and therefore it is not surprising that remotely these women are more at risk for hypertension, cardiovascular disease and stroke. Plasma volume has possibly a central role in the disease cascade, resulting in decreased cardiovascular reserve capacity. Furthermore a low plasma volume is found to be a strong predictor for recurrence of hypertensive complicated pregnancy. Adaptation, like in pregnancy, is for a large extent depending on the functioning of the venous compartment. In formerly preeclamptic women with low plasma volume is the venous compliance and capacitance decreased, furthermore there is sympathic hyperactivity. This combination reflects a decreased cardiovascular reserve capacity. These women with low plasma volume show a reduced ability to adapt their cardiovascular system to a new pregnancy.

It is known that physical exercise increases plasma volume in healthy adults, also arterial and both venous compliance and capacitance is improved by exercise. Since abnormal circulatory functions are common in formerly preeclamptic women, we want to study the effects of exercise in this specific group, and compare these results with women after an uneventful pregnancy. In preventive perspective it would be beneficial that also formerly preeclamptic women show a circulatory adaption to aerobic exercise, possibly they could improve their haemodynamic profile prior to their pregnancy

ELIGIBILITY:
Inclusion Criteria:

* patients: formerly preeclamptic women with history of preeclampsia (according to set criteria)
* controls: women with history of an uneventful pregnancy All women are examined at least 5 months postpartum;

Exclusion Criteria:

* pregnancy
* insulin dependant diabetes mellitus
* use of medication known to interfere with cardiovascular system
* incapability to cope with physical exercise
* auto immune disease

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Increase plasma volume | 3 months

SECONDARY OUTCOMES:
Venous Compliance | 3 months
Endothelial dysfunction | 3 months
Sympathetic resting activity | 3 months
Splanchnic blood flow | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spaanderman, Dr, Study Chair — Radboud University Medical Center Nijmegen
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Derived] Scholten RR, Hopman MT, Lotgering FK, Spaanderman ME. Aerobic Exercise Training in Formerly Preeclamptic Women: Effects on Venous Reserve. Hypertension. 2015 Nov;66(5):1058-65. doi: 10.1161/HYPERTENSIONAHA.115.05786. Epub 2015 Sep 8. PMID 26351026
- [Derived] Scholten RR, Spaanderman ME, Green DJ, Hopman MT, Thijssen DH. Retrograde shear rate in formerly preeclamptic and healthy women before and after exercise training: relationship with endothelial function. Am J Physiol Heart Circ Physiol. 2014 Aug 1;307(3):H418-25. doi: 10.1152/ajpheart.00128.2014. Epub 2014 Jun 6. PMID 24906915
- [Derived] Scholten RR, Thijssen DJ, Lotgering FK, Hopman MT, Spaanderman ME. Cardiovascular effects of aerobic exercise training in formerly preeclamptic women and healthy parous control subjects. Am J Obstet Gynecol. 2014 Nov;211(5):516.e1-516.e11. doi: 10.1016/j.ajog.2014.04.025. Epub 2014 Apr 23. PMID 24769012